CLINICAL TRIAL: NCT04218513
Title: An Experiment to Evaluate the Drug-drug Interaction of Formula Edaravone and Formula 2-Aminoethanesulfonic Acid in Compound Edaravone Injection
Brief Title: Drug-drug Interaction Study Between Edaravone and 2-Aminoethanesulfonic Acid in Compound Edaravone Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NJYK-CPEDRV-DDI
Record Dates: First submitted 2019-12-17; First posted 2020-01-06 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Drug-drug Interaction
Keywords: Drug-drug Interaction; Edaravone; 2-Aminoethanesulfonic Acid; Compound Edaravone Injection
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Intervention Model Description: Three-cycle crossover study
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compound Edaravone (Experimental): 30 mL (containing edaravone 30 mg and 2-aminoethanesulfonic acid 600 mg)
  Interventions: Drug: Compound Edaravone Injection
- Edaravone (Experimental): 30 mL (containing edaravone 30 mg)
  Interventions: Drug: Edaravone Injection
- 2-Aminoethanesulfonic Acid (Experimental): 30 mL (containing 2-aminoethanesulfonic acid 600 mg)
  Interventions: Drug: 2-Aminoethanesulfonic Acid Injection

INTERVENTIONS:
Drug: Compound Edaravone Injection — 30 min intravenous infusion
  Arms: Compound Edaravone
Drug: Edaravone Injection — 30 min intravenous infusion
  Arms: Edaravone
Drug: 2-Aminoethanesulfonic Acid Injection — 30 min intravenous infusion
  Arms: 2-Aminoethanesulfonic Acid

SUMMARY:
An experiment to evaluate the drug-drug interaction of formula edaravone and formula 2-aminoethanesulfonic acid in compound edaravone injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old (including upper and lower limits);
2. Weight ≥50 kg, body mass index (BMI) between 18-28 kg / m2 (including upper and lower limits);
3. Understand and sign the informed consent voluntarily, and volunteer to participate in this research.

Exclusion Criteria:

1. A history of diseases of the heart, liver, lung, kidney, digestive tract, blood, or neuropsychiatric system judged by the investigator as clinically significant;
2. A comprehensive physical examination, neurological examination, laboratory examination, ECG examination, or cognitive assessment indicates that the subject has an abnormality that the researcher has determined to be clinically significant;
3. Have taken any drug within two weeks before the study administration, and the researcher believes that this situation may affect the evaluation results of this study;
4. There is a history of food or drug allergy or allergies that the researcher judges to be clinically significant;
5. Those with positive results of serological examination (HBsAg, anti-HCV, anti-HIV, TP-Ab);
6. A history of alcohol or drug abuse that the investigator believes may affect the evaluation results of this study within one year before the study administration;
7. Cannot quit smoking or drinking during the study period or the carbon monoxide breath test> 7 ppm during the screening period CO breath test, so if the subject's CO breath is> 7ppm, but the urine cotinine test is negative, it means that the CO breath test result may be false positive, the subject can be enrolled;
8. As a subject who has participated in any drug clinical trial within 3 months before the first administration of the study;
9. Those who donated blood or blood products ≥400 mL or 2 units within three months of the study;
10. Do not agree to avoid the use of tobacco, alcohol or caffeinated beverages, or vigorous exercise, or other factors that affect drug absorption, distribution, metabolism, excretion, etc. during the 24 hours before and during the test;
11. Pregnant or lactating women, or those who tested positive for serum HCG before the test administration, or those who were unable or unwilling to take researcher-approved contraception during the study according to the researcher's instructions;
12. Subjects with poor compliance or unable to comply with the relevant provisions of the research protocol due to personal reasons, the investigator judges that the subjects are not suitable to participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Cmax of edaravone with and without coIntravenous with 2-Aminoethanesulfonic Acid | 24 hours
AUC0-t of edaravone with and without coIntravenous with 2-Aminoethanesulfonic Acid | 24 hours
AUC0-∞ of edaravone with and without coIntravenous with 2-Aminoethanesulfonic Acid | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China